CLINICAL TRIAL: NCT04960085
Title: Role of Echocardiography in the Assessment of Right Ventricular Function in the Pediatric Population With Valvular Pulmonary Stenosis After Percutaneous Balloon Pulmonary Valvuoplasty.
Brief Title: Role of Echocardiography in the Assessment of Right Ventricular Function in the Pediatric Population With Valvular Pulmonary Stenosis.
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Saad Abdelhafiz Abdelsalam, Egypt, Assuit, Assiut University
Other Study IDs: echo in RV function
Record Dates: First submitted 2021-07-02; First posted 2021-07-13 (Actual); Last update posted 2021-07-13 (Actual); Status verified 2021-07

CONDITIONS: Right Ventricular Dysfunction
MeSH Terms: conditions — Ventricular Dysfunction, Right | interventions — Echocardiography

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: echocardiography — philips IE33

SUMMARY:
Correct assessment of right ventricular function by transthoracic echocardiographic examination in pediatric patients with congenital valvular pulmonary stenosis after Percutaneous Balloon Pulmonary Valvuloplasty

DETAILED DESCRIPTION:
The right ventricle plays an important role in the morbidity and mortality of patients presenting with signs and symptoms of cardiopulmonary disease. However, the systematic assessment of right heart function is not uniformly carried out. This is due partly to the enormous attention given to the evaluation of the left heart, a lack of familiarity with ultrasound techniques that can be used in imaging the right heart, and a paucity of ultrasound studies providing normal reference values of right heart size and function. In patients with CHD, the right ventricle (RV) may function as either the sub-pulmonary or the systemic ventricle as in transposition of great arteries (TGA). CHD more commonly affecting the right heart includes atrial septal defects (ASD), Tetralogy of Fallot (TOF), pulmonary stenosis (PS), Ebstein anomaly, arrhythmogenic right ventricular cardiomyopathy (ARVC), and pulmonary valve atresia. In many of these patients, prevention of "irreversible" right heart failure (RHF) will require timely corrective surgery or when not possible, surgical palliation . Congenital pulmonary valve stenosis is a common congenital heart disease. Isolated pulmonary valve stenosis comprises 8-10% of all congenital heart disease . While surgical pulmonary valvotomy has been available as a treatment since 1956, it requires a median sternotomy, use of cardiopulmonary bypass, and post-surgical ICU admission with multi-day hospitalization. Recognizing the potential advantages of a less invasive approach, the first attempts at percutaneous catheter-based dilation of stenotic pulmonary valves were performed in the 1950s. As the technique was refined and catheter and balloon technology have advanced, the results of balloon pulmonary valvuloplasty have improved and the approach has become the standard of care for treating pulmonary valve stenosis

ELIGIBILITY:
Inclusion Criteria:

* All pediatric patients with congenital valvular pulmonary stenosis attending echocardiographic outpatient clinic of Assuit University children hospital aged from one month to18 years old

Exclusion Criteria:

Age less than one month and older than 18 years. Patients with infundibular and supravalvular pulmonary stenosis

Ages: 1 Month to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: pediatric patients with valvular pulmonary stenosis who will undergo trans cutaneous pulmonary valvuloplasty
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2021-07-02 (Estimated); Primary Completion 2022-07-02 (Estimated); Study Completion 2022-08-02 (Estimated)

PRIMARY OUTCOMES:
correlation between right ventricular dysfunction and severity of valvular pulmonary stenosis | baseline
  tissue Doppler of the right ventricle before and after trans cutaneous pulmonary valvuloplasty

REFERENCES:
- [Background] Pierpont ME, Basson CT, Benson DW Jr, Gelb BD, Giglia TM, Goldmuntz E, McGee G, Sable CA, Srivastava D, Webb CL; American Heart Association Congenital Cardiac Defects Committee, Council on Cardiovascular Disease in the Young. Genetic basis for congenital heart defects: current knowledge: a scientific statement from the American Heart Association Congenital Cardiac Defects Committee, Council on Cardiovascular Disease in the Young: endorsed by the American Academy of Pediatrics. Circulation. 2007 Jun 12;115(23):3015-38. doi: 10.1161/CIRCULATIONAHA.106.183056. Epub 2007 May 22. PMID 17519398
- [Background] Baumgartner H, Bonhoeffer P, De Groot NM, de Haan F, Deanfield JE, Galie N, Gatzoulis MA, Gohlke-Baerwolf C, Kaemmerer H, Kilner P, Meijboom F, Mulder BJ, Oechslin E, Oliver JM, Serraf A, Szatmari A, Thaulow E, Vouhe PR, Walma E; Task Force on the Management of Grown-up Congenital Heart Disease of the European Society of Cardiology (ESC); Association for European Paediatric Cardiology (AEPC); ESC Committee for Practice Guidelines (CPG). ESC Guidelines for the management of grown-up congenital heart disease (new version 2010). Eur Heart J. 2010 Dec;31(23):2915-57. doi: 10.1093/eurheartj/ehq249. Epub 2010 Aug 27. No abstract available. PMID 20801927
- [Background] Haddad F, Doyle R, Murphy DJ, Hunt SA. Right ventricular function in cardiovascular disease, part II: pathophysiology, clinical importance, and management of right ventricular failure. Circulation. 2008 Apr 1;117(13):1717-31. doi: 10.1161/CIRCULATIONAHA.107.653584. No abstract available. PMID 18378625
- [Background] Haddad F, Hunt SA, Rosenthal DN, Murphy DJ. Right ventricular function in cardiovascular disease, part I: Anatomy, physiology, aging, and functional assessment of the right ventricle. Circulation. 2008 Mar 18;117(11):1436-48. doi: 10.1161/CIRCULATIONAHA.107.653576. No abstract available. PMID 18347220
- [Background] Hornung TS, Bernard EJ, Jaeggi ET, Howman-Giles RB, Celermajer DS, Hawker RE. Myocardial perfusion defects and associated systemic ventricular dysfunction in congenitally corrected transposition of the great arteries. Heart. 1998 Oct;80(4):322-6. doi: 10.1136/hrt.80.4.322. PMID 9875104
- [Background] Hauser M, Bengel FM, Hager A, Kuehn A, Nekolla SG, Kaemmerer H, Schwaiger M, Hess J. Impaired myocardial blood flow and coronary flow reserve of the anatomical right systemic ventricle in patients with congenitally corrected transposition of the great arteries. Heart. 2003 Oct;89(10):1231-5. doi: 10.1136/heart.89.10.1231. PMID 12975428
- [Background] Davlouros PA, Niwa K, Webb G, Gatzoulis MA. The right ventricle in congenital heart disease. Heart. 2006 Apr;92 Suppl 1(Suppl 1):i27-38. doi: 10.1136/hrt.2005.077438. PMID 16543599
- [Background] Cheung MM, Smallhorn JF, Redington AN, Vogel M. The effects of changes in loading conditions and modulation of inotropic state on the myocardial performance index: comparison with conductance catheter measurements. Eur Heart J. 2004 Dec;25(24):2238-42. doi: 10.1016/j.ehj.2004.07.034. PMID 15589642
- [Background] Vogel M, Sponring J, Cullen S, Deanfield JE, Redington AN. Regional wall motion and abnormalities of electrical depolarization and repolarization in patients after surgical repair of tetralogy of Fallot. Circulation. 2001 Mar 27;103(12):1669-73. doi: 10.1161/01.cir.103.12.1669. PMID 11273995
- [Background] Vogel M, Schmidt MR, Kristiansen SB, Cheung M, White PA, Sorensen K, Redington AN. Validation of myocardial acceleration during isovolumic contraction as a novel noninvasive index of right ventricular contractility: comparison with ventricular pressure-volume relations in an animal model. Circulation. 2002 Apr 9;105(14):1693-9. doi: 10.1161/01.cir.0000013773.67850.ba. PMID 11940549
- [Background] Vogel M, Derrick G, White PA, Cullen S, Aichner H, Deanfield J, Redington AN. Systemic ventricular function in patients with transposition of the great arteries after atrial repair: a tissue Doppler and conductance catheter study. J Am Coll Cardiol. 2004 Jan 7;43(1):100-6. doi: 10.1016/j.jacc.2003.06.018. PMID 14715190